CLINICAL TRIAL: NCT04234178
Title: The Effects of Dural Puncture Epidural Versus Combined Spinal Epidural With Epidural Volume Extension Techniques on Birth Variables in Labor Analgesia
Brief Title: Dural Puncture Epidural Versus Combined Spinal Epidural With Epidural Volume Extension in Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammed E Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATATURKLABOR
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dural puncture epidural (Active Comparator): 2 µg/ml fentanyl + %0,125 bupivacaine (20 ml) to epidural
  Interventions: Drug: Epidural
- Combined spinal-epidural with epidural volume extension (Active Comparator): 10 µg fentanyl + 2 mg bupivacaine to intrathecal 7.4 ml saline volume to epidural
  Interventions: Drug: Intrathecal+Epidural

INTERVENTIONS:
Drug: Epidural — 2 µg/ml fentanyl + %0,125 bupivacaine (20 ml) to epidural
  Arms: Dural puncture epidural
Drug: Intrathecal+Epidural — 10 µg fentanyl + 2 mg bupivacaine to intrathecal 7.4 ml saline volume to epidural
  Arms: Combined spinal-epidural with epidural volume extension

SUMMARY:
Labor is the process where the cervix is prepared to allow the baby to pass from the uterine cavity to the outside world. In the ordinary course, it ends with spontaneous or instrumental vaginal delivery or cesarean section. Traditionally, the first stage in which the cervix is passively dilated in response to uterine contractions consists of the second stage in which the mother passes the baby through the vagina and the third stage, the exit of the placenta.

In the first stage of labor, pain is caused by uterine contractions and pressure on the cervix. Pain is transmitted through the T10-L2 spinal nerves and is felt in the abdominal wall, waist, hips, or thighs. In the second stage, pain from the vagina and perineum is added to uterine pain. This pain is transmitted by the pudendal nerves through the S2-4 nerve roots.

In this study, we aimed to investigate the effects of dural puncture epidural analgesia versus combined spinal-epidural analgesia with epidural volume extension on labor variables.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II parturients
* Pregnant patients in active labor
* active labor with cervical dilation < 5cm
* 37-42 weeks of gestational age
* Pregnant women between the ages of 18 and 45

Exclusion Criteria:

* Patients who do not want to participate voluntarily in the study
* Pregnant women outside the age range of 18 - 45
* Pregnants other than Nullipar
* Patients with allergic reactions to anesthesia and analgesia drugs to be used
* Severe systemic disease (kidney, liver, pulmonary, endocrine, cardiac)
* Gestational comorbidity (preeclampsia, eclampsia, diabetes mellitus, etc.)
* Substance abuse history
* Chronic pain history
* Psychiatric problems and communication difficulties
* BMI> 35 kg / m2
* Failure in neuraxial interventions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant patients
Enrollment: 60 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-07 (Actual)

PRIMARY OUTCOMES:
First Epidural top-up time | First 24 hours
  Time elapsed between the end of local anesthetic injection and the return of pain >4 on the NPRS.

SECONDARY OUTCOMES:
Sacral analgesia time | First 24 hours
  Blockade of the S2 dermatome
Performance time | First 24 hours
  interval between skin disinfection and epidural catheter fixation to the skin
Incidence of Side Effect | First 24 hours
  maternal motor block, hypotension, pruritis, headache and fetal bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed En Aydin, Principal Investigator — Ataturk University
Locations (2):
- Turkey (Türkiye) (2):
  - Ataturk University, Erzurum, Yakutiye
  - Erzurum Regional Training Research Hospital, Erzurum, Yakutiye

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Contreras F, Morales J, Bravo D, Layera S, Jara A, Riano C, Pizarro R, De La Fuente N, Aliste J, Finlayson RJ, Tran DQ. Dural puncture epidural analgesia for labor: a randomized comparison between 25-gauge and 27-gauge pencil point spinal needles. Reg Anesth Pain Med. 2019 May 22:rapm-2019-100608. doi: 10.1136/rapm-2019-100608. Online ahead of print. PMID 31118278
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Derived] Doymus O, Aydin ME, Bedir Z, Tor IH, Ejder Tekgunduz S, Doymus G, Celik EC, Ahiskalioglu A. Epidural volume extension versus dural puncture epidural analgesia for labor: A prospective randomized study. Medicine (Baltimore). 2025 Mar 7;104(10):e41691. doi: 10.1097/MD.0000000000041691. PMID 40068075